CLINICAL TRIAL: NCT06862830
Title: The Effectiveness of Virtual Reality in the Management of Procedural Anxiety and Pain in Children Suffering From Chronic Pathologies or Burn Injuries. Single-center Randomized Controlled Trial.
Brief Title: The Effectiveness of Virtual Reality in the Management of Procedural Anxiety and Pain in Children Suffering From Chronic Pathologies or Burn Injuries.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Biagio Nicolosi, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-PLS
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Anxiety; Chronic Disease; Pain
Keywords: Virtual Reality; Chronic pain; Paediatric; Chronic disease
MeSH Terms: conditions — Anxiety Disorders; Chronic Disease; Pain; Chronic Pain | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality video (Experimental)
  Interventions: Other: Virtual reality video
- Standard of care (No Intervention)

INTERVENTIONS:
Other: Virtual reality video — Virtual reality video: luna park, carousels, space, zoo, safari, dinosaurs, sightseeing, role-play
  Arms: Virtual reality video

SUMMARY:
Single-center, randomized, controlled clinical trial (RCT) to evaluate the efficacy of VR on pain and anxiety in children with chronic diseases undergoing painful procedures in an outpatient or day hospital setting

ELIGIBILITY:
Eligibility Criteria: Inclusion

The study population includes children who meet the following criteria:

1. Diagnosis of a chronic condition, aged 3 to 18 years, without visual impairments or cognitive deficits, and with a confirmed diagnosis of the condition.
2. Children receiving care in the wound care nursing clinic or Medical Day Hospital (DH) who require minimally invasive painful procedures.
3. Assent and informed consent provided by both the children and their parents.
4. Children with chronic conditions that do not inherently cause chronic pain, which could alter pain perception (e.g., rheumatoid arthritis, diabetic foot, muscular dystrophy).
5. Children able to understand and communicate in Italian or English.
6. Parents able to understand and communicate in Italian or English. Eligibility Criteria: Exclusion

Children with the following characteristics will be excluded from the study:

1. Chronic condition not yet diagnosed.
2. Use of eyeglasses, presence of amblyopia or monocular vision.
3. Chronic pain, which could distort pain perception during the procedure.
4. Use of analgesic therapy within the last 8 hours, which could bias data collection results (the only prohibited therapy in the study and a reason for exclusion).
5. Cognitive impairment preventing the proper use of assessment scales.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction in anxiety score | From recruitment to end of painful procedure
  Effectiveness of VR in reducing pain and anxiety in children undergoing painful procedures (blood draw, intramuscular injection, and wound dressing).
Percentage reduction in pain | From recruitment to end of painful procedure

SECONDARY OUTCOMES:
Percentage of reduction in parental anxiety | From recruitment to end of painful procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital IRCCS, Florence, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Nel presente studio, verranno condivisi i seguenti dati individuali dei pazienti (IPD) in forma anonimizzata e aggregata, garantendo il rispetto delle normative sulla privacy e sulla protezione dei dati personali:
  1. Dati Demografici e Clinici
     * Età del partecipante (fasce di età)
     * Genere
     * Patologia cronica principale
     * Eventuali comorbidità
     * Tipo di famiglia (monogenitoriale, entrambi i genitori, altro)
  2. Dati sulla Procedura e sull'Intervento
     * Tipo di procedura dolorosa eseguita (prelievo ematico, iniezione intramuscolare, medicazione)
     * Assegnazione del paziente al gruppo sperimentale (RV) o di controllo (cure standard)
  3. Dati sulla Valutazione dell'Ansia e del Dolore
     * Punteggi pre-procedurali di ansia anticipatoria valutati con:
     * M-YPAS (3-6 anni)
     * CAPS (6-17 anni e genitori)
     * Punteggi post-procedurali del dolore valutati con:
     * Wong-Baker Faces Scale (3-8 anni)
     * Numerical Rating Scale (NRS) (8-17 anni)
  4. Dati Statistici e di Outcome
     * Differenze nei p
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 01.09.2025 - 31.12.2025